CLINICAL TRIAL: NCT04666766
Title: Detecting Traumatic Intracranial Hemorrhage With Microwaves and Biomarkers: A Prospective Study Evaluating Ability of Microwave Scanning in Conjunction With Biomarkers to Diagnose Traumatic Intracranial Hemorrhage
Brief Title: Detecting Traumatic Intracranial Hemorrhage With Microwaves and Biomarkers
Acronym: MBI01
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Region Skane (Other)
Collaborators: Medfield Diagnostics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: MBI01
Record Dates: First submitted 2020-11-13; First posted 2020-12-14 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Brain Injuries, Traumatic; Biomarkers; Microwave Imaging
Keywords: Microwave Imaging
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: No results of the biomarker assays or microwave scans will be visible to the care givers or the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Traumatic intracranial hemorrhage (Active Comparator): Patients with traumatic intracranial hemorrhage diagnosed by Computerized Tomography of the head
  Interventions: Device: Microwave scanning of the head
- Trauma without traumatic intracranial hemorrhage (Active Comparator): Patients with trauma to the head but traumatic intracranial hemorrhage ruled out by Computerized tomography of the head
  Interventions: Device: Microwave scanning of the head
- Healthy age-matched volunteers (Active Comparator): Healthy age-matched volunteers with no previous trauma to the head within the past two weeks.
  Interventions: Device: Microwave scanning of the head

INTERVENTIONS:
Device: Microwave scanning of the head — A scan of the head will be performed with a microwave device to ascertain the likelihood of intracranial hemorrhage.
  Other Names: Assay of 9 different brain biomarkers

SUMMARY:
This study will evaluate if traumatic intracranial hemorrhage can be safely ruled out by using a microwave scanner (MD100) in conjunction with a combination of different brain biomarkers analyzed in serum.

DETAILED DESCRIPTION:
This is a prospective, open, multicentre trial that will enrol patients presenting to the Emergency Department (ED) because of isolated head trauma or head trauma as part of a multi trauma. Microwave scanning characteristics and biomarkers in patients with traumatic intracranial haemorrhage (TICH) (Group A) will be compared to patients with head trauma that do not have TICH (Group B). All adult patients with trauma to the head will be eligible for inclusion if a medical professional has evaluated the risk of spine injury. After additional physical examination, control of inclusion- and exclusion criteria and after informed consent has been acquired, the microwave measurement and blood sampling will be performed. Before enrolment in the study, and in the acute phase, one of the investigators or a member of the investigator staff must explain verbally the implications of study participation to the patient, and the patient is asked to give a verbal consent. As soon as is practically possible after the acute phase of the disease, the patient will sign and personally date the informed consent form. In cases where the patient is not capable to read and/or sign the informed consent, due to disability, an independent witness shall be present throughout the process of reading the written informed consent and any other information aloud and explained to the prospective patient. As an independent witness, healthcare professionals who are not responsible or in any way involved in the patient's care or treatment are accepted. The independent witness can sign on the behalf of the patient in the presence of the patient and the Investigator. More details of the informed consent procedure are described in this Clinical Investigation Plan, section 6.3.

The microwave measurement will take less than five minutes (the duration of the actual measurement is about 1,5 min and will not interfere with the patient's standard of care). The Research Nurse or the Investigator documents all patient clinical trial information in the eCRF.

Safety and usability will be evaluated throughout the trial, and a safety follow-up will be performed by the Research Nurse or Investigator approximately 24 hours after the measurement procedure.

During the data processing phase of study, the result of the microwave measurement will be compared to the result of the biomarkers, CT examination and the patient's final diagnosis. As a control group, approximately 50 demographically matched healthy volunteers (Group C) will be asked to participate in the trial. The trial will provide knowledge of the predictive value of microwave measurement and biomarkers for the diagnosis of intracranial haemorrhages in the acute TBI phase.

ELIGIBILITY:
Inclusion Criteria (groups A and B):

* Verbal Informed Consent in the acute phase.
* Signed Informed Consent Form after the acute phase. On behalf of the patient, independent witness signed informed consent (in cases where the patient is unable to sign).
* Acute trauma patient with suspected head injury
* Time from injury to measurement procedure not longer than 8 hours 15 min
* Head CT prescribed by treating physician
* Patient is ≥ 18 years of age
* Patient is deemed clinically stable

Exclusion Criteria (groups A and B):

* Patient has suspected cervical spine fracture, per the Investigator's judgement
* Patient has by CT confirmed cervical spine fracture
* Patient has confirmed skull fracture with risk for dislocation.
* Patient has a shunt or other foreign object implanted intracranially (if known by medical records)
* Patient has agraffes or other metal parts, thick bandage (>1cm), or other foreign materials attached to the head that are deemed to interfere with the diagnostic procedure.
* Patient diagnosed with a condition associated with risk of poor protocol compliance
* The measurement procedure is deemed to interfere with the standard of care
* Other condition or symptoms preventing the patient from entering the trial, per the investigator´s judgment

Inclusion Criteria (Group C):

* Patient is ≥ 18 years of age
* Signed informed consent

Exclusion Criteria (Group C):

• Previous stroke or other diagnosed and/or treated brain injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-01-10 (Estimated); Study Completion 2026-01-12 (Estimated)

PRIMARY OUTCOMES:
Ability to detect intracranial hemorrhage | 3.5 years
  The ability of the device MD100, with and without brain biomarkers (Aβ40, Aβ42, GFAP, H-FABP, S100B, NF-L, NSE, UCH-L1 and IL-10) to detect traumatic intracranial haemorrhage, as measured by the area under the receiver operating characteristics curve.

SECONDARY OUTCOMES:
Estimating anatomic position of intracranial hemorrhage | 3.5 years
  The accuracy for estimating the position of intracranial hemorrhage with microwave data.
Estimating volume of intracranial hemorrhage | 3.5 years
  The accuracy for estimating the volume of intracranial hemorrhage with microwave data.
Adverse events of microwave scan | 3.5 years
  Any adverse events occurring within 24 hours of microwave scan

CONTACTS AND LOCATIONS:
Overall Officials: Tomas J Vedin, MD, PhD, Principal Investigator — Region Skåne and Lund University
Locations (1):
- Helsingborg General Hospital, Helsingborg, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vedin T, Bergenfeldt H, Holmstrom E, Lundager-Forberg J, Edelhamre M. Microwave scan and brain biomarkers to rule out intracranial hemorrhage: study protocol of a planned prospective study (MBI01). Eur J Trauma Emerg Surg. 2022 Apr;48(2):1335-1342. doi: 10.1007/s00068-021-01671-7. Epub 2021 May 4. PMID 33944977